CLINICAL TRIAL: NCT04327284
Title: Immediate vs Delayed Placement of Straumann BLX Implants in Molar Extraction Sockets
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Research cancelled
Sponsor: Ahmad Kutkut (Other)
Collaborators: Straumann USA (Unknown)
Responsible Party: Sponsor-Investigator, Ahmad Kutkut, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 55344
Record Dates: First submitted 2020-03-26; First posted 2020-03-31 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Immediate Placement of Straumann BLX Implants in Molar Extraction Sockets
Keywords: Immediate; Molar; Extraction; Sockets; Bone Graft; Dental Implant

STUDY DESIGN:
Intervention Model Description: This study will be a single site, randomized, controlled, prospective, and parallel arms study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- test group (Experimental): The test group will receive immediate molar implant placement in fresh extraction socket with nonocclusal loading immediate provisionalization (Straumann BLX 6.5mm).
  Interventions: Device: Immediate placement non-occlusal loading molar implant (Straumann BLX 6.5mm)
- Control group (Active Comparator): The control group will receive delayed molar implant placement at least 12 weeks post molar extraction with nonocclusal loading immediate provisionalization (Straumann BLX 5.0mm).
  Interventions: Device: Delayed placement non-occlusal loading molar implant (Straumann BLX 5.0mm)

INTERVENTIONS:
Device: Immediate placement non-occlusal loading molar implant (Straumann BLX 6.5mm) — At the screening visit, potential subjects will be informed about the protocol and all questions related to the study will be answered. Medical and dental histories will be reviewed and physical evaluations will be performed in order to rule out local or systemic factors that would compromise the outcome of the study. A detailed extra and intra oral examination will be performed. Appropriate radiographic imaging studies will be obtained prior to the surgical visit (per the protocol of the University of Kentucky, College of Dentistry) including CBCT and intraoral scans for treatment planning implant through Straumann Guided Surgery workflow.
  The duration of the present study is 1 year including the baseline or surgical visit, 2-weeks postoperative visit, 12-weeks baseline for control group and postoperative evaluations at 3, and 12 months.
  Arms: test group
Device: Delayed placement non-occlusal loading molar implant (Straumann BLX 5.0mm) — At the screening visit, potential subjects will be informed about the protocol and all questions related to the study will be answered. Medical and dental histories will be reviewed and physical evaluations will be performed in order to rule out local or systemic factors that would compromise the outcome of the study. A detailed extra and intra oral examination will be performed. Appropriate radiographic imaging studies will be obtained prior to the surgical visit (per the protocol of the University of Kentucky, College of Dentistry) including CBCT and intraoral scans for treatment planning implant through Straumann Guided Surgery workflow.
  The duration of the present study is 1 year including the baseline or surgical visit, 2-weeks postoperative visit, 12-weeks baseline for control group and postoperative evaluations at 3, and 12 months.
  Arms: Control group

SUMMARY:
The aim of this study is to clinically and radiographically compare the success and survival of implants immediately placed in molar fresh extraction socket to delayed implant placement at least 12 weeks post molar extraction. The secondary aim is to evaluate the peri-implant tissue response around implants with immediate vs. delayed placement.

DETAILED DESCRIPTION:
Study Population To be included in the study, the subjects must be 22 years of age or older and in good general health. They must have at least one nonrestorable more indicated for extraction and immediate or delayed implant placement. Subjects who are unable to undergo oral surgery procedures, smokers, and women who are (or become) pregnant (or are breastfeeding) will be excluded from this study. Additionally, subjects with bone infections or compromised health that may affect the ability of the patients' tissues to heal (e.g., uncontrolled diabetes, bisphosphonate use, current glucocorticoid use) will not be included in this clinical study.

15 implants in each group are necessary to provide 90% power with a type I error of 0.05. Each subject will be randomly assigned into one of two treatment groups:

Test Group (n=15):

The test group will receive immediate molar implant placement in fresh extraction socket with nonocclusal loading immediate provisionalization (Straumann BLX 6.5mm).

Control Group (n=15):

The control group will receive delayed molar implant placement at least 12 weeks post molar extraction with nonocclusal loading immediate provisionalization (Straumann BLX 5.0mm).

Subject Recruitment Methods and Privacy:

Subjects who seek implant treatment in University of Kentucky, College of Dentistry clinics. Implant clinics is referral base clinic. Once a subject is referred to extract a nonrestorable molar tooth and be replaced with an implant, potential subjects will be informed with the study. If subjects decide to be part of the study, informed consent will be signed prior to screening visit.

Informed Consent Process:

The research study will be conducted at the facilities of University of Kentucky, College of Dentistry after approval by the Institutional Review Board. All members of the research team received training in human subject protection. After each patient has been given verbal and written information describing the nature of the study, informed consent will be obtained before he or she can enter the study. A copy of the consent form will be given to the patient and another retained by the investigator. Patients will not be screened until an informed consent has been obtained.

ELIGIBILITY:
Inclusion Criteria:

* 22 years of age or older
* good general health.
* at least one nonrestorable more indicated for extraction and immediate or delayed implant placement

Exclusion Criteria:

* undergo oral surgery procedures
* smokers
* women who are (or become) pregnant (or are breastfeeding)
* subjects with bone infections or compromised health that may affect the ability of the patients' tissues to heal (e.g., uncontrolled diabetes, bisphosphonate use, current glucocorticoid use)

Ages: 22 Years to 78 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Clinical Examination: Implant Success and Failure Criteria | 12 months
  Implant success is defined by clinical and radiographic parameters. The success criteria for the implants will be (1) no radiolucency around the implant, (2) no mobility, and (3) no suppuration, pain, or ongoing pathologic process. Implants that do not meet the above criteria fall under the implant failure category. Success rate percentage will be based on clinical and radiographic assessment per implant site.
Radiographic Examination | 12 months
  Regional Cone Beam CT scan imaging for implant sites will be made for research purposes at baseline after implant placement, and 12 months follow up visits. These images are the only way to provide 3 dimensional view of bone around implants (Mesial-Distal, Buccal-Lingual). Marginal bone level changes will be recorded on the mid-mesial, mid-distal, mid-labial, and mid-lingual sites for each implant from the reference line (RL) of the implant platform immediately after implant placement and 12 months follow up visits. All measurements will be made utilizing a coDiagnostiX software used at University of Kentucky College of Dentistry. Marginal bone changes around implants for each site (i.e., Mesial, Distal, Buccal, and Lingual) will be digitally analyzed using the software and statistically analyzed and compared between groups utilizing SPSS software.
Osstell Value Assessment | 12 months
  Osstell® RFA (Resonance Frequency Analysis) values will be recorded immediately after implant placement, 3 months, and 12 months follow up visits to report implant stability during the healing time. RFA values for each implant will be statistically analyzed and compared between and within groups utilizing SPSS software.
3D Printed Models Assessment | 12 months
  3D printed models will be generated from intraoral scan prior to baseline extraction visit and 3, 12 months follow up. Volumetric changes will be measured and analyzed digitally with compare software.
Photographic Documentation | 12 months
  Photographic documentation will be made using a digital camera for each visit to clinically evaluate the peri-implant tissue healing response around implants with immediate vs. early placements.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad KutKut, DDS, MS, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No